CLINICAL TRIAL: NCT06185829
Title: Evaluating the Benefit of Hypnoanalgesia Versus Neuroleptanalgesia During Hand Surgery
Acronym: HYPNOMAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Vivactis M2Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-A00880-45
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Hand Surgery

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, randomized, open label study with two parallel groups of patients.
  Maximum duration of patient participation = 3 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual neuroleptanalgesic treatment (Active Comparator): Usual neuroleptanalgesic treatment Hypnovel (1 mg if weight < 60 kg, 1.5 mg if weight between 60 and 80 kg, 2 mg if weight > 80 kg)
  Interventions: Drug: Neuroleptanalgesic treatment
- Hypnoanalgesia (Experimental): Patients in this group will begin their hypnoanalgesia session with a nurse trained in hypnotherapy. Various methods commonly used in hypnosis (VAKOG, dissociation, diversion, metaphors, etc.) will be selected based on the patient, their personality, their expectations, and their degree of suggestibility.
  Interventions: Other: Hypnoanalgesia

INTERVENTIONS:
Drug: Neuroleptanalgesic treatment — Usual neuroleptanalgesic treatment Hypnovel and Locoregional anesthesia
  Other Names: Hypnovel
  Arms: Usual neuroleptanalgesic treatment
Other: Hypnoanalgesia — Hypnoanalgesia and Locoregional anesthesia
  Arms: Hypnoanalgesia

SUMMARY:
This is a single-center, prospective, randomized, open-label study of two parallel groups of patients undergoing hand surgery:

Group 1: locoregional anesthesia + neuroleptanalgesia Group 2: locoregional anesthesia + hypnoanalgesia Therapeutic benefit is based on VAS assessment of intraoperative anxiety.

DETAILED DESCRIPTION:
In a population of patients undergoing hand surgery and divided into two groups according to the anesthesia protocol administered in addition to locoregional anesthesia by truncal block:

Group 1: neuroleptanalgesia Group 2: hypnoanalgesia Primary objective The main objective of the study is to compare changes in preoperative anxiety between the two groups, between two measurements taken preoperatively (before anxiety management) and at the end of surgery. This level will be evaluated using a VAS rated from 0 to 10.

Secondary objectives

Comparing groups:

* Intraoperative pain
* Total duration of surgical procedure, ICU stay and hospitalization
* Amount of additional sedative treatment administered during surgery
* Post-operative pain
* Patient satisfaction
* Intraoperative and immediate postoperative adverse events

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 80,
* Patient who has read and signed the consent form for participation in the study after a reflection period (approximately 15 minutes).
* Patient applying for outpatient hand surgery under LRA, such as upper limb trunk blocks (flexor teno synovectomy or endoscopic carpal tunnel surgery).
* Patient requiring sedation associated with locoregional anaesthesia

Exclusion Criteria:

* Contraindication to locoregional anaesthesia or to one of the sedatives used in the protocol
* Pregnant or breastfeeding patient or woman of childbearing age without highly effective contraception for the duration of the study (surgically sterile, intrauterine device (> 14 days), hormonal contraception (same dose and formulation for at least 6 months), sexual abstinence. Women of childbearing age, i.e. fertile, are considered to be women after menarche and until they become post-menopausal, unless they are permanently infertile or have undergone surgical sterilisation. A post-menopausal state is defined as the absence of menstruation for 12 months without any other medical cause.
* Patient under court protection, guardianship or curatorship
* Patient not affiliated to the French social security system
* Patients unable to understand informed information and/or give written informed consent: dementia, psychosis, disturbed consciousness, non-French-speaking patients, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
VAS anxiety score | Day 2
  Changes in VAS anxiety score between preoperative and intraoperative assessment.
  Anxiety will be assessed on a visual analog scale measuring 10 cm (with 0 = no stress - 10 = major stress) and by administering the APAIS scale.

SECONDARY OUTCOMES:
Pain intensity assessment | Day 0
  Pain intensity will be assessed using a simple numerical scale (ENS) graduated from 0 (no pain) to 10 (worst pain imaginable).
Pain intensity assessment | Day 2
  Pain intensity will be assessed using a simple numerical scale (ENS) graduated from 0 (no pain) to 10 (worst pain imaginable).
Overall patient satisfaction | Day 0
  Overall patient satisfaction will be assessed using a simple numerical scale (ENS) graduated from 0 (not at all satisfied) to 10 (completely satisfied).
Overall patient satisfaction | Day 2
  Overall patient satisfaction will be assessed using a simple numerical scale (ENS) graduated from 0 (not at all satisfied) to 10 (completely satisfied).
Treatment Safety | Day 2
  The safety will be assessed by collecting data on adverse events occurring during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Mélanie FROMENTIN, MD, Principal Investigator — Hôpital Privé Paul d'Egine
Locations (1):
- Hôpital Privé Paul d'Egine, Champigny-sur-Marne, France

IPD SHARING:
Plan to Share IPD: No